CLINICAL TRIAL: NCT00602485
Title: The Effect of Action Control Based Interventions on Adherence to Prescribed Exercise and Diet Regimens for Patients Completing a Cardiac Rehabilitation Program Intervetnion on
Brief Title: The Effect of Action Control Based Intervention on Adherence After Cardiac Rehabilitaiton
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Summa Health System (Other)
Responsible Party: Donna Waechter, Ph.D., Summa Health System
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R07026
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Heart Failure
Keywords: adherence, cardiac rehabilitation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Action Control Education — 30 minute educational intervnetion

SUMMARY:
This will be a pilot study of the effect of an Action Control-based intervention (ACBI) on adherence to prescribed diet and exercise programs after cardaic rehabilitation. The purposes of this study are to:

1. determine if an ACBI has an effect on adherence to prescribed home exercise and diet regimens for individuals 6 weeks after participating in a cardiac rehabilitation program
2. examine whether there is a difference in response to the ACBI between state-oriented individuals and action-oriented individuals.
3. test the interaction effect between action-orientation disposition and the intervention.

DETAILED DESCRIPTION:
Patients with cardiac problems are burdened with complex lifestyle changes involving medication, diet and exercise. Non-adherence to prescribed treatment protocols is a major contributor to morbidity and mortality for these indiviudals. Rehabbilitation programs provide the necessary education and supervision needed to promote health, however, non-adherence occurs even for those indiviudals with appropriate resources and motivation. Most of the research up to this point deals with preparing indiviudals to be adherent. Action Control theory is focused on the mental processes that occur between the time an individual makes a decision to adhere and the moment when the appropriate activty either occurs or does not occur.

This interventions tudy will compare rates of adherece between indivudals who receive an action control based educational intervention and those who do not.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be a convenience sample of English literate men and women over the age of 21 enrolled in a cardiac rehabilitation program and accessible by phone for follow-up. All participants are referred to rehabilitation by their physician. Being enrolled in the program indicates the participants have experienced a serious cardiac event, either myocardial infarction and/or coronary surgery

Exclusion Criteria:

* Non-English literate, uner teh age of 21

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-06; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
self-report adherence to exercise and diet prescriptions | 6 weeks post cardaic rehabilitation

SECONDARY OUTCOMES:
action control orientaiton based on adherence | 6 weeks post cardaic rehabilitaiotn

CONTACTS AND LOCATIONS:
Overall Officials: Carrie J Scotto, PhD, Principal Investigator — Summa Health System
Locations (1):
- Summa Health System, Akron, Ohio, United States